CLINICAL TRIAL: NCT06127745
Title: A Prospective Study to Assess the Safety and Performance of the Discure Technologies System for the Treatment of Early to Moderate Degenerative Disc Disease (DDD).
Brief Title: Discure Technologies Feasibility Study for DDD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Discure Technologies Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN 002
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Degenerative Disc Disease; Chronic Low-back Pain; Discogenic Pain
Keywords: Discure System
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Intervention Model Description: All enrolled participants will be treated with the Discure System
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Discure System (Experimental): All participants enrolled in the study will be treated with the Discure system
  Interventions: Device: Discure System

INTERVENTIONS:
Device: Discure System — All subjects enrolled into the study will be implanted with the Discure System in a minimally invasive procedure.

SUMMARY:
The objective of this study is to evaluate the safety and performance of the Discure System therapy in subjects with early to moderate degeneration of the disc (DDD).

DETAILED DESCRIPTION:
A prospective, interventional, multi-center, single arm, open label, feasibility study. The study is designed to evaluate the safety and performance of the Discure System in the treatment of chronic low back pain (with or without radicular pain) of discogenic origin with early to moderate degeneration of the disc (DDD) in levels L1-2 to L5-S1, as confirmed by history and radiographic studies and/or discography, who failed conservative treatment of 12 weeks in duration.

Subjects will be followed at 1,3-, and 6-months post procedure. The primary endpoint will be assessed at the 6-month follow-up visit.

The study will enroll up to 20 subjects at up to 8 sites.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is ≥ 22 and ≤75 years of age.
2. If female of childbearing potential, participant is non-pregnant, non-nursing, and agrees to use highly effective methods of contraception for a minimum of 24 months post-treatment.
3. Participant has a documented diagnosis of early to moderate degenerative disc disease, confirmed by medical history, physical and neurological examination.
4. Participant has a discogenic mechanical Low Back Pain (LBP) of an intervertebral disc/s from L1 to S1, based on the following (participant must meet all the listed conditions):

   1. Chronic mechanical (axial) low back pain for at least 6 months
   2. Have failed 3 months of conservative back pain care
   3. Change from normal disc morphology of the index disc as defined on magnetic resonance imaging (MRI) and Xray evaluation must show the following:

      * Single level or up to two symptomatic (causing chronic LBP) discs from L1 to S1
      * A modified Pfirrmann score of 3, 4, 5 or 6 on magnetic resonance imaging (MRI) at the index disc/s.
      * Modic Grade II changes or less on MRI at the index disc.
      * With or without contained disc protrusion, with no nerve compression, at the index disc on MRI.
5. Low back pain of at least 40mm and not more than 90mm of 100mm on low back pain visual analogue scale (VAS) (average pain over 7 days diary)
6. Low back pain predominant over leg pain on a 100mm VAS scale
7. Oswestry disability index (ODI) score of at least 30 and no more than 90 on a 100- point scale.
8. Participant has the ability to comply with the instructions for use of the Discure System.
9. Participant is suitable for Discure system surgery as determined by the implanting physician prior to inclusion.
10. Participant is deemed to be neuro-psycho-socially appropriate for implantation. therapies based on a physician's assessment.

Exclusion Criteria:

1. BMI > 35
2. Back Pain characteristics:

   * Any surgical correction procedure for scoliosis at any time, or a current clinical diagnosis of scoliosis
   * Lumbar spine stenosis, as defined by an anterior-posterior diameter of the spinal canal of <10mm in participants with lower extremity pain
   * Neurological deficit possibly associated with the back pain (e.g. foot drop)
   * Back pain due to pelvic or visceral reasons (e.g.: endometriosis or fibroids) or infection (e.g.: post herpetic neuralgia)
   * Back pain due to damage to the spinal cord or adjacent structures (e.g., arachnoiditis or syringomyelia)
   * Pathology seen on MRI, other than DDD, that is clearly identified and is likely the cause of the Chronic Low Back Pain (CLBP) that is surgical.
   * Back pain due to other causes, such as vascular (e.g., aortic aneurysm and dissection), GI, GYU, oncological etc.
3. Source of pain is the sacroiliac joint or facet joint as determined by the Investigator.
4. Any prior diagnosis of lumbar vertebral compression fracture, lumbar pars fracture, or lumbar annular tear with disc protrusion of the target operative disc, that is surgical.
5. Participant has lumbar spondylitis or other undifferentiated spondyloarthropathy at the target disc.
6. Participant has had previous lumbar spine surgery at level L1-2 to L5-S1
7. Participant has had previous disc invasive treatment procedures, into the target disc/s, except for contrast media-discography performed at least 2 weeks prior to study enrollment.
8. Participant has symptomatic involvement of more than two lumbar discs or more than two lumbar discs that satisfy the radiographic profile defined in the Inclusion Criteria
9. Participant has current infection at the planned procedure site, active systemic infection, or current or prior history of lumbar spinal infection (i.e., discitis, septic arthritis, epidural abscess)
10. Participant is at higher risk for post-surgical infection (e.g., taking immunosuppressants, has a severe infection or a history of serious infection)
11. Participant has an active malignancy or tumor.
12. Participant has had significant systemic disease, such as unstable angina, autoimmune disease, rheumatoid arthritis, diabetes mellitus-insulin dependent, or muscular dystrophy.
13. Participant has a congenital or acquired coagulopathy or thrombocytopenia.
14. Participant is currently taking anticoagulant, antineoplastic, antiplatelet, or thrombocytopenia inducing medications (except for aspirin or nonsteroidal anti- inflammatory drugs [NSAIDS])
15. Participant has concomitant conditions requiring daily oral steroid usage for more than 30 days in the preceding 90 days before enrollment.
16. Participant has an uncontrolled psychiatric condition: bipolar disorder, post-traumatic stress disorder (PTSD) or uncontrolled anxiety/depression and/or require new or changed anti-depressants or anti-psychotic medications within 3 months of enrollment.
17. Participant has evidence of substance/ alcohol abuse that would potentially interfere with the participant's participation in the study within 3 months prior to enrollment.
18. Participant has or requires non-MRI compatible devices, such as an implantable electronic defibrillator, pacemaker, or has other contraindication to MRI scanning or cannot tolerate MRI scanning. Participants who are expected to require a defibrillator or pacemaker within the first 6 months of the study should be excluded.
19. Compensation injuries or ongoing litigation regarding back pain/ injury, or financial or other incentives to remain impaired.
20. Participant is currently enrolled in or plans to enroll in any concurrent drug, and/or biological, and/or device study while participating in this study.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Safety- Serious Adverse Events | 6 months
  Assessment of serious device and/or procedure related adverse events (SAE) in all participants.
Performance | 6 months
  The change from baseline in functional disability on the Oswestry Disability Index (ODI) measured from 0 (minimal disability) to 100 (maximal disability) OR The mean change of low back pain as measured by a 0 (no pain)-100 mm (worst pain) Visual Analogue Scale (VAS) 7-day diary from baseline to primary endpoint visit.

SECONDARY OUTCOMES:
Patient Satisfaction | 6 months
  The change in patient satisfaction as measured by Patient Global Impression of Change (PGIC) from baseline to 6 months visit.
Participant Quality of Life | 6 months
  The change in Quality of Life as measured by the European Quality of Life Five 5 Dimension (EQ-5D) from baseline to 6 months visit, scored from 100 ('the best health state you can imagine') to 0 ('the worst health you can imagine').
Pain Medication | 6 months
  Pain medication usage reduction

IPD SHARING:
Plan to Share IPD: No